CLINICAL TRIAL: NCT03921255
Title: Developing Interpretation Training for Modifying Thought Action Fusion Associated With Obsessive-compulsive Symptoms
Brief Title: Cognitive Bias Modification for Thought-Action Fusion
Acronym: TAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Milwaukee (Other)
Responsible Party: Principal Investigator, Han Joo Lee, Associate Professor, University of Wisconsin, Milwaukee
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAF Extended
Record Dates: First submitted 2019-03-10; First posted 2019-04-19 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Thought-Action Fusion; Cognitive Bias Modification; Interpretation Training; Stress Management Psychoeducation
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: Three training groups, assessed at pre-training, post-training, and follow-up.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are randomized to one of three training conditions. The randomized training assignment is unknown to the participant and assessor by using code names for the training conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TAF Incongruent (TAF-INC) (Active Comparator): Active condition (TAF-INC) cognitive bias modification for interpretations (CBM-I), incorporates an obsessional thought meant to elicit either moral or likelihood TAF, followed by a sentence incongruent to TAF bias and meant to reduce the impact of the previous statement. Before moving on, participants must fill-in and correctly solve a key word important in the interpretation of the sentence. Participants then must correctly solve a short yes/no comprehension question to ensure understanding of the scenario.
  Interventions: Other: Cognitive Bias Modification
- TAF Congruent (TAF-CON) (Placebo Comparator): Maintenance/Control condition (TAF-CON) CBM-I, differs in that participants are provided with a sentence congruent with TAF bias. Again, participants were only able to move on when they correctly solved the key word and the accompanying yes/no comprehension question.
  Interventions: Other: Cognitive Bias Modification
- Stress Management Psychoeducation (Placebo Comparator): In the stress management psychoeducation (SMP) psychoeducation about stress and stress management are provided, similar in length to the obsessional thought and interpretations presented in the TAF-INC and TAF-CON. Like the other conditions there is a key word to solve, and participants were only able to move on when they correctly solved the key word and the accompanying yes/no comprehension question.
  Interventions: Other: Cognitive Bias Modification

INTERVENTIONS:
Other: Cognitive Bias Modification — There is support that CBM-I may work through the process of cognitive restructuring, and specifically, threat reappraisal. Threat appraisal is a tendency to overestimate the likelihood of harm (i.e., likelihood bias) and/or the negative consequences of anticipated harm (i.e., Clark & Beck, 2010), producing avoidance, thus interfering with effectively reappraising threat, thereby creating a vicious cycle (Beck et al., 1985; Clark & Beck, 2010). CBM-I procedures ensure that an interpretation bias is triggered by the ambiguous scenarios, and participants are then guided to solve the key word in accordance with a healthy response (Grey & Mathews, 2000). The observed effects of CBM-I may stem from active generation of benign or positive meanings in response to ambiguous situations, where threats were previously interpreted (Beadel et al., 2014).
  Other Names: Interpretation Training

SUMMARY:
An important cognitive bias in many emotional disorders, particularly obsessive-compulsive disorder (OCD), is thought-action fusion (TAF). TAF describes the bias to interpret the presence of unwanted mental intrusions as morally equivalent to acting on them (TAF-M), and/or increasing the likelihood of the feared consequence occurring to either oneself (TAF-LS) or others (TAF-LO). The present study is designed to test the feasibility of a single session computerized cognitive bias modification for interpretations (CBM-I) to reduce TAF among individuals who reported obsessional intrusions. Participants will be randomized to (a) the TAF-incongruent condition (TAF-INC), designed to decrease TAF linked to obsessional thoughts, to (b) the TAF-congruent condition (TAF-CON), designed to render TAF-like interpretation of obsessional thoughts unchallenged, or to (c) a Stress Management Psychoeducation (SMP) condition, designed to provide information about stress reduction, but not target TAF directly.

DETAILED DESCRIPTION:
Individuals who display at least mild obsessional and TAF symptoms will be invited to the current study. Participants will be randomized to one of the three interpretation training conditions: an TAF-INC, TAF-CON, or SMP. Before and after the training, participants will complete some self-report questionnaires and clinician administered measures. The computerized training will provide statements intended to activate the mechanisms involved in thought-action-fusion (TAF), which will almost always produce a negative outcome interpretation. It is hypothesized that through TAF-INC participants will learn alternative, more neutral, ways of interpreting the thoughts and lower the subject's TAF. The TAF-CON condition will receive the same statements as TAF-INC, but TAF-CON is designed to leave the interpretation of the scenarios unchallenged. The study will also include another comparison condition, SMP, to test if TAF-INC outperforms not only TAF-CON, but also stress reduction techniques provided in empirically supported psychological treatment. The SMP training will be similar in procedure and structure to the other two conditions, but it will provide psychoeducation about stress and stress management techniques.

ELIGIBILITY:
Inclusion Criteria:

* UWM undergraduates who were at least 18 years old who (i) score of at least 1 [A Little (Distressed or Bothered)] on the OCI-R obsessing subscale, and (ii) at least one TAFS item scored 3 (Agree) or 4 (Agree Strongly) were be eligible to participate in the study. A score of 1 or higher on the obsessing subscale of the OCI-R indicates the presence of obsessional intrusions, and was used as a cutoff in previous research (Siwiec et al., 2017). A score of 3 or above on an item of the TAFS indicates the participant agrees with and holds some pronounced TAF bias.

Exclusion Criteria:

* Individuals whose primary language is not English will not be included in the study. Assessment and training programs are all written in English (we are not able to present a version in another language) - it is important for participants to understand subtlety of slightly varying vignettes in the training program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-04-10 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Thought-Action Fusion Scale (TAFS) across Pre-training, Post-training, and 1-Month follow-up | Pre-training, post-training (same day as pre-training), 1-Month Follow-up
  The Thought-Action-Fusion Scale (TAFS; Shafran et al., 1996) is a 19-item measure which assesses the degree to which importance and responsibility is lent to a variety of intrusive and distressing thoughts containing moral and likelihood themes. The measure uses a 5-point scale ranging from 0 (Disagree Strongly), to 4 (Agree Strongly). There are no cutoff scores but higher TAFS scores are indicative of higher rates of TAF cognitions (Shafran et al., 1996). In student and community samples the three-scale model (TAF-M, TAF-LS, TAF-LO) has displayed moderate to strong association between the scales (r=.25 - .69; Abramowitz et al., 2003; Bailey et al., 2014; Coles, Mennin, & Heimberg, 2001; Rassin, Merkelbach et al., 2001).

SECONDARY OUTCOMES:
Change in Primary Obsession Evaluation of TAF Scale (POETS) across Pre-training, Post-training, and 1-Month follow-up | Pre-training, Post-training (same day as pre-training), 1-Month Follow-up
  The Primary Obsession Evaluation of TAF Scale (POETS; Siwiec et al., 2017) is designed to assess the participant's TAF emotional and cognitive reactions toward a specific (primary) obsessional intrusion. A study clinician helps identify their primary obsessive thought using the Y-BOCS Obsession Checklist. The POETS uses a 7-point scale from 0 (Not Distressing at All), to 6 (Extremely Distressing), and incorporates 3 domains (5 questions each): (1) General Emotional Reactions, (2) Moral TAF, and (3) Likelihood TAF. The general emotional reaction domain gauges discomfort with the presence of the thought, the moral domain gauges the moral implications of the thought, and the likelihood domain gauges the belief to which the event will occur because of the thought.
Change in Revised Obsessional Intrusions Inventory - Distress (ROII-Distress) across Pre-training, Post-training, and 1-Month follow-up | Pre-training, Post-training (same day as pre-training), 1-Month Follow-up
  The Revised Obsessional Intrusions Inventory - Distress (ROII-Distress) is a 52-item self-report measure, modified (Siwiec et al., 2017) from the original ROII (Purdon & Clark, 1993, 1994), to assess how distressing various intrusive thoughts, images, and impulses would be to the participant in the event of their intrusion. The measure uses a 7-point scale from 0 (Not Distressing), to 6 (Extremely Distressing). Unlike the original ROII, the ROII-Distress does not use a time frame as the obsessive thoughts, images, or impulses may not have occurred yet, but asks instead of distress if the thought were to occur. In consideration of heterogeneity in obsessional intrusions across individuals, we computed an idiographic distress index, consisting of the 10-highest endorsed ROII-Distress items for each participant at pre-training.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Siwiec, M.S., Principal Investigator — University of Wisconsin, Milwaukee
Locations (1):
- UWM Anxiety Disorders Laboratory, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UWM Anxiety Disorders Lab Website — https://sites.google.com/site/uwmanxiety/
- See also: UWM SONA Portal to Prescreen Information — http://uwm.edu/psychology/undergraduate/participate-sona/